CLINICAL TRIAL: NCT05153109
Title: Reliabilty and Validity of a Diagnostic Interview for Parents of Babies and Preschoolers
Brief Title: Reliabilty and Validity of a Diagnostic Interview for Parents of Babies and Preescholers
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Ruth von Brachel, Principal Invertigator, Ruhr University of Bochum
Other Study IDs: 553
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Psychological Disease
Keywords: clinical interview

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Community sample: Participants will be recruited from families in Bochum who take part in experiments and studies at the department of delevopmental psychology at the Ruhr-University. The department of developmental psychology organizes a panel every year inviting all parents of newborn babies in Bochum to register if they want to participate in research.
- Clinical sample: Participants will be recruited from families in Bochum and Munich who seek treatment in the outpatient treatment centers at both sites. Both study sites offer special counselling for parents who experience difficulties with a child from zero to five years of age.

SUMMARY:
The Kleinkind-DIPS (Diagnostisches Interview bei psychischen Störungen für Kleinkinder) is a structured interview to assess a variety of the most frequent psychological problems in babies and preschoolers, e.g. feeding or sleeping problems, anxiety disorders. It is administered by a trained clinician with one of the primary carers. In this study, its acceptance, reliability and validity will be tested in a clinical and non-clinical sample.

DETAILED DESCRIPTION:
The Kleinkind- DIPS (Diagnostisches Interview bei psychischen Störungen für Kleinkinder) is a structured interview to assess a variety of the most frequent psychological of the most frequent psychological problems in babies and preschoolers, e.g. feeding or sleeping problems, anxiety disorders. It is administered by a trained clinician with one of the primary carers. In this study, its acceptance, reliability and validity will be tested in a clinical and non-clinical sample. Parts of the interview are adapted from the Kinder-DIPS, for which information on acceptance, reliability and validity are available. The aim of the present study is to test the interviews acceptance, reliability and validity in both a clinical and a non-clinical sample.

ELIGIBILITY:
Inclusion Criteria: sufficient knowledge of the German language -

Exclusion Criteria:

-

Ages: 0 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All parents who have a child in the according age group.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Kleinkind-DIPS | within one week of the other measures
  structured interview for parents of preschoolers

SECONDARY OUTCOMES:
Fragebogen zum Schreien, Füttern, Schlafen (SFS) | within one week of the other measures; only for parents of children aged 18 months or younger
  Questionnaire assessing feeding, sleeping and crying in young infants, three subscales: feeding problems, sleep problems, coregulation; scores (means) ranging from 1-4, higher scores indicate more problems
Depression Anxiety Stress Scale (DASS-21) | within one week of the other measures;
  Questionnaire assessing depression, anxiety and stress of the parents, higher scores indicate higher stress or psychopathology; depression scores range from 0-28; stress scores 0-34, anxiety 0-20;
Strengths and Difficulties Questionnaire (SDQ) | within one week of the other measures; only for parents of children aged 18 months or older
  Questionnaire assessing internalizing and externalizing problems in children; 5 sub scales of which 4 capture problems (e.g. emotional difficulties, conduct problems) and one scale which captures prosocial behaviour; For each of the 5 scales the score can range from 0 to 10 with higher scores indicating more problems and more prosocial behaviour
Parental sense of control (PSCO) | within one week of the other measures;
  Questionnaire assessing self-efficacy and sense of control of the parents; Two subsacles: efficacy and satisfaction; means between 1-6. A higher score indicates a higher parenting sense of competency.

OTHER OUTCOMES:
Acceptance of the Interview | within one week after being interviewed
  Questionnaire assessing parents perception of the interview, 10 Items assessing 5 positive and 5 negative attitudes towards the interview, higher scores indicate higher endorsement. One additional item assessing global satisfaction with the interview on a scale from 0-100, higher scores indicate higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Schneider, Phd, Study Director — Ruhr University of Bochum
Locations (2):
- Germany (2):
  - Ludwig Maximilian University of Munich, Munich, Bavaria
  - Ruhr-University, Bochum, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No
we cannot share individual participant data due to data protection constrictions